CLINICAL TRIAL: NCT01187368
Title: Prospective Multi-Center Randomized Study for Evaluating the EVAHEART®2 Left Ventricular Assist System: the COMPETENCE Trial
Brief Title: Prospective Multi-Center Randomized Study for Evaluating the EVAHEART®2 Left Ventricular Assist System
Acronym: COMPETENCE
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Subject recruitment is temporarily on hold due to ongoing device modification.
Sponsor: Evaheart, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 020-1601-001-P01
Record Dates: First submitted 2010-08-19; First posted 2010-08-24 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure
Keywords: Heart failure; LVAS; LVAD; Bridge-to-transplant; Continuous flow pump; Destination therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Three-hundred and ninety-nine (399) subjects will be enrolled and randomized in a 2:1 assignment to receive EVA2 or the comparator device, HeartMate 3.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Evaheart LVAS (EVA2) (Experimental): The objective of the study is to evaluate the safety and effectiveness of the EVA2 by demonstrating non-inferiority to commercially approved LVADs when used for the treatment of refractory NYHA Class III with dyspnea upon mild physical activity or Class IV heart failure.
  Interventions: Device: EVAHEART Left Ventricular Assist System (LVAS)
- HeartMate 3 (HM3) (Active Comparator): The objective of the study is to evaluate the safety and effectiveness of the EVA2 by demonstrating non-inferiority to commercially approved LVADs when used for the treatment of refractory NYHA Class III with dyspnea upon mild physical activity or Class IV heart failure.
  Interventions: Device: HeartMate 3

INTERVENTIONS:
Device: EVAHEART Left Ventricular Assist System (LVAS) — Three-hundred and ninety-nine (399) subjects will be enrolled and randomized in a 2:1 assignment to receive EVA2 or the comparator device, HeartMate 3.
  Other Names: EVA2
  Arms: Evaheart LVAS (EVA2)
Device: HeartMate 3 — Three-hundred and ninety-nine (399) subjects will be enrolled and randomized in a 2:1 assignment to receive EVA2 or the comparator device, HeartMate 3.
  Other Names: HM3
  Arms: HeartMate 3 (HM3)

SUMMARY:
This is a prospective, multi-center, unblinded, randomized, controlled, and non-inferiority study comparing the EVA2 LVAS to the most recent magnetically levitated centrifugal LVAS (HM3 LVAS).

DETAILED DESCRIPTION:
Adult (>18 years old), advanced heart failure NYHA Class III with dyspnea upon mild physical activity or Class IV patients who are refractory to advanced heart failure management and meet study Inclusion/Exclusion criteria will be enrolled.

The objective of the study is to evaluate the safety and effectiveness of the EVA2 by demonstrating non-inferiority to commercially approved LVADs when used for the treatment of refractory advanced heart failure.

Subjects will be followed for 6 months (short-term cohort) and 24 months (long-term cohort) after EVA2/HM3 LVAS implantation or until outcome events of transplantation, explantation, death or withdrawal, whichever occurs first. Whereas subjects experiencing the outcome events of "Severe RHF" and "Disabling stroke" will remain in study follow-up.

ELIGIBILITY:
Inclusion Criteria:

The following is a list of general inclusion criteria:

* Age ≥ 18 years
* Left Ventricular Ejection Fraction (LVEF) < 30%
* NYHA Class III with dyspnea upon mild physical activity or Class IV heart failure
* Inotrope dependent OR Cardiac Index (CI) < 2.2 L/min/m2, while not on inotropes
* Patient is able to provide written informed consent
* More detailed inclusion criteria information is noted in the study protocol

Exclusion Criteria:

1. Etiology of heart failure due to or associated with uncorrected thyroid disease, obstructive cardiomyopathy, pericardial disease, amyloidosis, or restrictive cardiomyopathy
2. Technical obstacles which pose an inordinately high surgical risk
3. Existence of ongoing mechanical circulatory support (MCS) other than IABP and Impella 5.0 or 5.5
4. Ongoing Impella (5.0 or 5.5) presenting related clinical sign (i.e. hematuria) and elevated LDH equal or greater than 600 IU/L.
5. Positive pregnancy test if of childbearing potential
6. Presence of mechanical aortic cardiac valve that will not be either converted to a bioprosthesis
7. History of any organ transplant
8. Platelet count <100,000/mL
9. Psychiatric disease/disorder, irreversible cognitive dysfunction or psychosocial issues
10. History of confirmed, untreated abdominal aortic aneurysm (AAA) > 5 cm in diameter within 6 months of enrollment
11. Presence of an active, uncontrolled infection
12. Intolerance to anticoagulant or antiplatelet therapies or any other peri/postoperative therapy that the investigator will require based upon the patient's health status
13. Presence of remarkable pre-defined end-organ dysfunction.
14. Patient has moderate to severe aortic insufficiency without plans for correction during pump implant
15. Low albumin - removed from recent exclusion criteria
16. Planned Bi-VAD support prior to enrollment
17. Patient has known hypo- or hyper coagulable state such as disseminated intravascular coagulation and heparin induced thrombocytopenia (HIT)
18. Participation in any other clinical investigation that is likely to confound study results or affect the study
19. Any condition other than heart failure that could limit survival to less than 24 months
20. Patients refusing blood transfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Estimated)
Dates: Start 2020-03-31 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Short-Term Primary Endpoint | 6 months
  Survival to cardiac transplant or device explant for recovery free from disabling stroke (Modified Rankin Score > 3) or pre-defined severe Right Heart Failure at 6 months after implantation of the originally implanted device
Long-Term Primary Endpoint | 24 months
  Survival to cardiac transplant or device explant for recovery free from disabling stroke (Modified Rankin Score > 3) or pre-defined severe Right Heart Failure at 24 months after implantation of the originally implanted device

SECONDARY OUTCOMES:
Change in KCCQ and EuroQol | Baseline versus POD 30, 90, 180, 360 and every 180 days
Change in 6-minute walk test | Baseline versus POD 30, 90, 180, 360 and every 180 days
NYHA functional class | Baseline versus POD 30, 90, 180, 360, and every 180 days
Frequency and incidence of all re-operations | Discharge after implant through transplant or explant for recovery.
Frequency and incidence of all rehospitalizations | Discharge after implant through transplant or explant for recovery.
Incidence of adverse events, serious adverse events and UADEs | Implant through transplant or explant for recovery (+60 days or discharge) or 180 days on device; then duration of device support, up to 360 days (approximate)
  Peri-operative complications and any failure to successfully implant the device.
  All adverse events occurring during the acute and chronic phase of the study (frequency, severity, duration, sequelae and relationship to device).
  All adverse events occurring during the extension phase (frequency, severity, duration, sequelae and relationship to device).
Incidence of all device failures and device malfunctions | Implant through transplant or explant for recovery (+60 days or discharge) or 180 days on device; then duration of device support, up to 360 days(approximate)
Post-transplant or post-explant survival | Up to 30 days post-transplant or post-explant

OTHER OUTCOMES:
Powered Secondary Endpoint: GI bleeding | 24 months
  Documented mucosal (GI tract and/or nasopharynx) bleeding, requiring blood transfusion (backed red blood cells) or hemoglobin drop (>2 g/dL) without another identifiable source of bleeding AND meet one or more of the following:
  * Identified mucosal bleeding by endoscope
  * Appearance of overt melena, hematochezia, hematemesis, epistaxis
  * Occult bleeding as evidenced by hemoccult-positive stool (2 consecutive testing to avoid false positive)

CONTACTS AND LOCATIONS:
Overall Officials: Tadashi Motomura, MD, PhD, Study Director — Evaheart, Inc.
Locations (12):
- United States (12):
  - UF Health Shands Hospital, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - St. Vincent Hospital Indianapolis, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - The Christ Hospital, Cincinnati, Ohio
  - Penn State Health Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Baylor Scott and White, Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Methodist Hospital - San Antonio, San Antonio, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - University of Wisconsin-Madison, Madison, Wisconsin